CLINICAL TRIAL: NCT03263468
Title: Revascularization StrategIes for ST Elevation Myocardial Infarction Trial
Acronym: ASSIST-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-254
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: ST Elevation Myocardial Infarction; Coronary Stenting; Primary Angioplasty
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Same sitting complete revascularization (Experimental): After treatment of the IRA, subjects will undergo PCI of all suitable significant non-IRA lesions (≥70% by visual assessment or FFR<0.80 in 50-70% lesions with vessel diameter >2mm).
  Interventions: Procedure: Same sitting PCI with complete revascularization
- Staged non-IRA PCI (Active Comparator): Only the IRA will be intervened upon during the index primary PCI procedure. Staging of the non-IRA lesions will be performed 48 hours to 45 days after the primary PCI procedure. All suitable non-IRA lesions (≥70% by visual assessment or FFR<0.80 in 50-70% lesions with vessel diameter >2mm) will be treated with PCI irrespective of whether there are clinical symptoms or evidence of ischemia.
  Interventions: Procedure: Staged PCI with complete revsacularization >48 hours pf primary PCI

INTERVENTIONS:
Procedure: Same sitting PCI with complete revascularization — revascualrization of the non IRA (infarct related artery) of > 2.0 mm by coronary angioplasty/stenting at the time of primary PCI
  Arms: Same sitting complete revascularization
Procedure: Staged PCI with complete revsacularization >48 hours pf primary PCI — revascualrization of the non IRA (infarct related artery) of > 2.0 mm by coronary angioplasty/stenting >48 hours to 45 days post primary PCI
  Arms: Staged non-IRA PCI

SUMMARY:
This study is being conducted in patients with a major heart attack caused by a blocked artery undergoing Percutaneous Coronary Intervention (PCI) to open up the blockage. Up to 50% of people with an heart attack are found to have one or more additional narrowings that did not cause the heart attack. At present the best way to manage these additional blockages is not known. Many cardiologist recommend opening these blockages at at a later time after the heart attack. The present study is examining if PCI of all blockages at the same time as the PCI for the artery that caused the major heart attack (SS-PCI) will reduce the amount of heart damage compared to performing PCI of additional blockages 2-45 days later (IRA-PCI). Clinical follow up will be completed at 3, 12 and 24 months to determine heart function and monitor adverse events.

ELIGIBILITY:
Inclusion Criteria:

* ST elevation myocardial infarction evidenced by new ST elevation at the J point in at least 2 contiguous leads of ≥ 2 mm (0.2mV) in men or ≥ 1.5mm (0.15mV) in women in leads V2-V3 and/or ≥ 1mm (0.1mV) in other contiguous chest leads or limb leads.
* MVD as evidenced by > one significant (>70% by visual assessment or FFR < 0.80 for 50-70% stenosis) stenosis in the non-IRA >2mm in diameter.
* Successful IRA-PCI with <30% residual angiographic stenosis and TIMI III flow
* Written informed consent

Exclusion Criteria:

* Age ≤ 18 years
* Prior coronary artery bypass graft (CABG) surgery
* Administration of thrombolytic therapy.
* Hemodynamic instability as evidenced by SBP<90 mmHg, Killip class ≥3, and/or need for inotropes/vasopressors.
* Known renal insufficiency (estimated GFR < 30 ml/min/1.73m2)
* Non-IRA stenosis is a chronic total occlusion (CTO)
* Plan by treating physician to treat non-IRA stenosis with coronary artery bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3520 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse clinical events | 90 days
  Composite of all-cause mortality, myocardial infarction, heart failure and unplanned revascularization

SECONDARY OUTCOMES:
Major bleeding | 90 days
Stroke | 90 days
Contrast nephropathy | 90 days
Major vascular complication | 90 days
EQ-5D quality of life assessment | 90 days
Incremental Cost-Effectiveness Ratio (ICER) | 90 days
Myocardial infarction | 90 days
Heart failure | 90 days
All cause mortality | 90 days
Unplanned revascularization | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Bagai, MD, Principal Investigator — Unity Health Toronto; Asim Cheema, MD, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: Undecided